CLINICAL TRIAL: NCT05599347
Title: Pre-treatment With Azithromycin to Reduce Immunogenicity to Anti-Tumor Necrosis Factor-α Agents in Patients With Crohn's Disease
Brief Title: Pre-treatment With Azithromycin to Reduce Immunogenicity to to Anti-TNF Agents in Patients With Crohn's Disease
Acronym: AZITRATIM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Haggai Bar-Yoseph MD, Principal investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0432-22-RMB
Record Dates: First submitted 2022-09-14; First posted 2022-10-31 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Crohn's Disease Relapse; Biological Substance; Adverse Effect
Keywords: Crohn's disease; infliximab; adalimumab; azithromycin; immunogenicity
MeSH Terms: conditions — Crohn Disease | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: All consenting adults that fulfil the inclusion criteria will be randomized in a 1:1 ratio and allocated to the azithromycin or placebo arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin (Experimental): 5-day consecutive treatment with oral azithromycin 500 mg once daily
  Interventions: Drug: Azithromycin Pill
- Control (Placebo Comparator): 5-day consecutive oral placebo once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Azithromycin Pill — Tablet - 500 mg azithromycin (as dihydrate)
  Arms: Azithromycin
Other: Placebo — Placebo tablet identical in shape and appearance to the azithromycin tablet used in the treatment arm
  Arms: Control

SUMMARY:
This is a randomized placebo-controlled trial in Crohn's disease patients before initiation of anti-tumor necrosis factor-α (anti-TNF) therapy that aims to test the effect of a pre-treatment short course of azithromycin therapy on immunogenicity

DETAILED DESCRIPTION:
Anti-TNF agents are considered the mainstay of therapy for patients with inflammatory bowel diseases (IBD). Still, its efficacy is hampered by the development of anti-drug antibodies (ADA), which lead to non-responsiveness to this medication. A combination with immunosuppressive agents is currently utilized to reduce ADA development but is accompanied by an increased risk of side effects (i.e. malignancy and infections). The investigators have recently found an epidemiologic link between prior antibiotic use and the development of ADA, and shown an antibiotic-specific effect on ADA development in a mouse model. Macrolide antibiotics were specifically associated with ADA prevention and led to increased durability of the treatment. Since the microbiome has been associated with the response to anti-TNF therapy, the investigators hypothesize that microbial manipulation with azithromycin prior to the initiation of anti-TNF therapy will lower ADA development. the investigators propose a randomized controlled study to test our hypothesis and compare it to matched historical cohorts with available clinical and serological data. The primary outcome will be ADA development at 1 year of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent prior to any study procedures and willing and able to attend all study visits, comply with the study procedures, read and write in order to complete questionnaires, and be able to complete the study period.
* Aged 18 to 80 years of age, inclusive, at the time of signing the informed consent.
* Diagnosis of CD with an onset of symptoms for a minimum of 3 months prior to Screening as determined by the investigator based on clinical history, exclusion of infectious causes, and characteristic endoscopic and histologic findings.
* Prior decision of starting infliximab or adalimumab therapy (including biosimilar drugs).
* Thiopurine and corticosteroid co-therapy will be permitted.

Exclusion Criteria:

* Inclusion in another interventional study
* Patients who cannot provide informed consent and do not have a legal guardian
* Patients with perianal involvement who are expected to require antibiotic therapy for their disease
* Patients on chronic antibiotic therapy due to any cause
* Patients with ongoing fluid collection/abscess either internal or perianal
* Known history of allergy to the study intervention formulation or any of its excipients or components of the delivery device
* Prolonged QTc interval or conditions leading to additional risk for QT prolongation
* Chronic kidney disease stage 5 (GFR < 10)
* Crohn's Disease complication requiring surgical treatment
* Planned/ongoing methotrexate co-therapy
* Fecal microbiota transplantation within 8 weeks prior to randomization
* Participant has any disorder that, in the opinion of the investigator, may compromise the ability to participate in the study
* Pregnancy
* Patients who received azithromycin therapy in the previous year (we will not exclude prior use of other antibiotic therapy)
* Patients who received any antibiotic treatment within 4 weeks prior to randomization
* Re-induction of the same anti-TNF medication
* Patients who are on chronic therapy which cannot be withheld in one of these medications: colchicine, phenytoin, and digoxin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Anti-drug antibody development | 1 year after the initiation of therapy
  Percent of patients developing anti-drug antibodies defined as measurable antibodies using an anti-lambda ELISA assay

SECONDARY OUTCOMES:
Sustained corticosteroid-free clinical remission | At both 3 months and a 1 year after the initiation of therapy
  Crohn's Disease Activity Index (CDAI) ≤150 without systemic corticosteroid therapy
Clinical response | 1 year after the initiation of therapy
  A reduction in CDAI of at least 100 points from baseline.
Sustained corticosteroid-free biochemical remission | at both 6 months and a 1 year after the initiation of therapy
  C-reactive protein (CRP) ≤1.5 upper limit of normal, or fecal calprotectin ≤ 250 mg/kg
Treatment durability | at both 6 months and a 1 year after the initiation of therapy
  Persistent administration of infliximab or adalimumab for 1 year. A 16-week or more interval between infliximab injections, or an 8-week or more interval between adalimumab injections will be considered as treatment cessation. Change in anti-TNF regimen at 26 and 52 weeks defined as increased dosing or decreased dosing interval
Anti-TNF drug levels | At 6 weeks, 26 weeks and a 1 year after the initiation of therapy
  Levels at various timepoints
Early anti-drug antibody development | At 6 weeks, 26 weeks and a 1 year after the initiation of therapy
  Percent of patients developing anti-drug antibodies defined as measurable antibodies using an anti-lambda ELISA assay
PRO-2 remission at Week 52 | 1 year after the initiation of therapy
  - Patient reported outcome (PRO-2) remission at Week 52 (defined as an abdominal pain [AP] mean daily score at or below 1 [AP≤1] AND a stool frequency [SF] mean daily score at or below 3 [SF≤3], and no worsening of AP or SF from baseline).
Sustained corticosteroid-free PRO-2 clinical remission | At both 14 and a 1 year after the initiation of therapy
  The rate of sustained corticosteroid-free PRO-2 clinical remission at both 14 and 52 weeks, defined as AP≤1 and SF≤3. The rate of clinical response at 14 weeks, defined as a reduction in CDAI of at least 100 points from baseline
Addition of immunomodulator treatment | At any time during the study
  The rate of addition of immunomodulator treatment defined as at least one dose of thiopurines or methotrexate
Immunomodulator treatment termination | At 14 weeks and not restarting by 1 year after the initiation of therapy
  The rate of immunomodulator treatment termination. Termination will be defined in patient treated with azathioprine or 6MP at randomization, as being stopped after at least 14 weeks and not restarting by 52 weeks
Endoscopic improvement | At 26 weeks
  Endoscopic improvement defined as a reduction of ≥50% decrement from baseline in SES-CD score
Endoscopic remission | At 26 and 52 weeks
  Endoscopic remission defined as SES-CD ≤4

CONTACTS AND LOCATIONS:
Locations (9):
- Israel (9):
  - Soroka University Medical Center, Beersheba
  - Bnei Zion, Haifa
  - Carmel Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Shaare Zedek, Jerusalem
  - Zvulun, Kiryat Bialik
  - Rabin Medical Center, Petah Tikva

REFERENCES:
- [Result] Gorelik Y, Freilich S, Gerassy-Vainberg S, Pressman S, Friss C, Blatt A, Focht G, Weisband YL, Greenfeld S, Kariv R, Lederman N, Dotan I, Geva-Zatorsky N, Shen-Orr SS, Kashi Y, Chowers Y; IIRN. Antibiotic use differentially affects the risk of anti-drug antibody formation during anti-TNFalpha therapy in inflammatory bowel disease patients: a report from the epi-IIRN. Gut. 2022 Feb;71(2):287-295. doi: 10.1136/gutjnl-2021-325185. Epub 2021 Aug 3. PMID 34344783